CLINICAL TRIAL: NCT05782491
Title: Rapid Progression of Care in Cardiogenic Shock - Awake Surgical Placement of the Impella 5.5 Using Regional Anesthesia
Brief Title: Awake Axillary Impella 5.5 Placement - A Feasibility Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research decided not to pursue.
Sponsor: University of Pennsylvania (Other)
Collaborators: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 852788; 77327727 (Other Grant/Funding Number: Abiomed)
Record Dates: First submitted 2023-02-24; First posted 2023-03-23 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Cardiogenic Shock
Keywords: Impella 5.5; Cardiogenic shock; PECS II; Interscalene; Superficial Cervical; regional anesthesia
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Cervical Plexus Block

STUDY DESIGN:
Intervention Model Description: 10 patients in cardiogenic shock listed for Impella 5.5 placement
Masking Description: No blinding in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patient in cardiogenic shock listed for Impella 5.5 placement who meets study inclusion criteria
  Interventions: Procedure: Interscalene Block; Procedure: PECS II Block; Procedure: Superficial Cervical Plexus Block

INTERVENTIONS:
Procedure: Interscalene Block — It is an ultrasound guided brachial plexus nerve block at roots/trunks used to anesthetize the shoulder and upper arm. Goal is to spread local anesthetic around superior and middle trunks of brachial plexus, between the anterior and middle scalene muscles.
  Other Names: Peripheral nerve block
Procedure: PECS II Block — PECS II block is comprised of two separate fascial plane blocks to anesthetize anterolateral chest wall using an ultrasound guided injection between the pectoralis major muscle and pectoralis minor muscle at third rib and a second ultrasound guided injection between pectoralis minor and serratus anterior. The goal is a high volume hydro dissection of the two fascial planes to anesthetize anterolateral chest wall and axilla.
  Other Names: Pectoral Block; Peripheral nerve block; Fascial plane block
Procedure: Superficial Cervical Plexus Block — This block is a superficial injection to the deep cervical fascia between the investing layer of the deep cervical fascia and the prevertebral fascia in the neck. This block provides anesthesia of the skin of the anterolateral neck and the ante-auricular and retro-auricular areas, as well as the skin overlying and immediately inferior to the clavicle on the chest wall. This is an ultrasound guided injection with the goal of placing the needle tip in the fascial layer underneath the SCM adjacent to the cervical plexus, which is contained within the tissue space between the Cervical fascia and posterior sheath of the SCM.
  Other Names: Cervical plexus block; Peripheral nerve block

SUMMARY:
The Abiomed Impella 5.5 is a surgically placed temporary mechanical support device used in patients in cardiogenic shock. The investigators propose using regional anesthesia (3 separate peripheral nerve blocks) to facilitate Impella 5.5 placement, a procedure which has traditionally been performed under a general anesthetic.

Regional anesthesia is a proven and widely used technique to facilitate upper extremity vascular surgery cases (i.e. arteriovenous fistula creation). The investigators believe that employing these blocks in conjunction with intravenous sedation or monitored anesthesia care (MAC anesthesia) - a technique used in all types of cases, even in sick hearts during thranscatheter aortic valve replacements (TAVR) - will avoid the need increased doses of medications to support the blood pressure and cardiac output, avoid the need for post operative mechanical ventilation and intravenous sedation, and speed up the time to participating in physical therapy, time to heart transplant/durable mechanical support/recovery, and time to hospital discharge.

DETAILED DESCRIPTION:
General anesthesia places patients who are in cardiogenic shock at risk for life threatening hemodynamic compromise due to the anesthetic and positive pressure ventilation, and confers the need for mechanical ventilation and sedation post operatively.

Our hypothesis is that by utilizing regional anesthesia, anesthesiologists can facilitate surgical Impella placement with less risk of cardiovascular collapse with a faster road to recovery. By avoiding endotracheal intubation and concomitant heavy sedation both in the operating room and ICU, these patients will avoid worsening deconditioning and ICU delirium, with less days to physical therapy, ambulation, and recovery as compared to patients who undergo general anesthesia and remain ventilated in the ICU after their Impella placement.

Patients scheduled for Impella 5.5 placement will be screened by a specific set of inclusion/exclusion criteria for potential participation in the study. If they consent, they will receive three commonly used upper extremity nerve blocks (Interscalene, PECS II, and superficial cervical plexus nerve blocks) and receive only intravenous sedation during the procedure.

ELIGIBILITY:
Inclusion Criteria:

Baseline Criteria:

* Agrees to procedure
* Excellent ultrasound images for nerve blocks
* Excellent ultrasound images for trans thoracic echo
* Age <60, BMI <30
* Non hostile neck
* Evaluation of CT amenable to easy surgical access for Impella placement

Meets criteria for MAC sedation:

* Able to lay relatively flat comfortably
* Able to understand and cooperate with procedures
* Easy airway (Mallampati I - II, prior grade 1-2 airway)
* Low risk of airway obstruction
* No high baseline oxygen requirement (over 6L/min)

Meets criteria for regional anesthesia:

* Patient agrees to nerve block
* No active areas of infection around the block site
* No history of nerve damage or deficits in the area of the proposed nerve block
* No contralateral diaphragmatic paralysis or phrenic nerve palsy

Exclusion Criteria:

* Does not wish to have MAC
* Does not wish to have Regional Anesthesia
* BMI > 30
* Poor U/S windows for block or TTE
* Active infection over block area
* High Oxygen Requirement >6L NC
* Known or anticipated difficult airway
* Unable to lay flat comfortably Unable to cooperate or follow instructions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Success of Using Regional Anesthesia for Impella 5.5 Placement | Day of procedure (1 day)
  Number of patients that successfully undergo Impella 5.5. placement with the regional anesthesia protocol

SECONDARY OUTCOMES:
Time to participation in physical therapy | 6 weeks
  Time from end of operation to getting out of bed or involving in physical therapy sessions
Time to destination therapy | 6 weeks
  Time to decision of heart transplant, ventricular assist device, or recovery
Sedation requirement | 1 week
  Total dose of sedatives required post operatively
Pain medication requirement | 1 week
  Total dose of pain medication required post operatively
Patient pain scores post operatively | 3 days
  The Numeric Pain Rating Scale score on post operative evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Asad Usman, MD, MPH, Principal Investigator — University of Pennsylvania; Marisa Cevasco, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No